CLINICAL TRIAL: NCT03717909
Title: A Pivotal, International, Randomised, Double-blind, Efficacy and Safety Trial of Sodium Valproate, in Paediatric and Adult Patients With Wolfram Syndrome
Brief Title: Efficacy and Safety Trial of Sodium Valproate, in Paediatric and Adult Patients With Wolfram Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: RG_16_211
Record Dates: First submitted 2018-10-11; First posted 2018-10-24 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Wolfram Syndrome
Keywords: Wolfram Syndrome; Treat Wolfram; Sodium valproate
MeSH Terms: conditions — Wolfram Syndrome | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Sodium Valproate 200Mg E/C Tablet (active treatment)
  Interventions: Drug: Sodium Valproate 200Mg E/C Tablet
- Control Group (Placebo Comparator): Sodium Valproate matched placebo (inactive treatment)
  Interventions: Drug: Sodium Valproate matched placebo

INTERVENTIONS:
Drug: Sodium Valproate 200Mg E/C Tablet — Treatment with twice-daily oral tablet(s)
  Other Names: Sodium Valproate
  Arms: Experimental Group
Drug: Sodium Valproate matched placebo — Treatment with twice-daily oral 200mg tablet(s)
  Other Names: Placebo
  Arms: Control Group

SUMMARY:
This trial aims to investigate the efficacy, safety and tolerability of sodium valproate in the treatment of patients with Wolfram syndrome. 70 paediatric and adult patients were initially planned to be randomised 2:1 to receive either sodium valproate or placebo at 6 international centres. 63 patients were recruited when a decision was made to stop the study recruitment in November 2022.

DETAILED DESCRIPTION:
This phase II clinical trial is planned as a randomised, double-blind, placebo-controlled 3 year intervention Trial in 70 patients with Classical Wolfram Syndrome aged 6 years and over. The primary outcome of the Trial is considered to be clinically relevant and of sufficient magnitude to be beneficial, as a successful Trial outcome will mean that patients will retain a clinically useful degree of visual acuity and it will decline at a slower rate than in the untreated patients. The MRI Pons Volume change has been shown to correlate with changes in the Wolfram Unified Rating Scale.

Patients will be randomised to balance the individual differences across the treatment and placebo groups, therefore reducing the potential for extraneous bias. This will ensure that the treatment effect can be established without the need to account for confounding factors. The value of a placebo arm adds robustness to the Trial by removing the potential for bias from both the investigator and patient perspectives.

Investigators will be blinded to the results of the assessments. Certain assessments will be performed by subspecialists (such as ophthalmologists and neurologists), with the Principal Investigator prevented from having access to the results. This subspecialist-led treatment is in line with the current multi-disciplinary management of these patients and will not result in patients being denied access to effective treatment.

Patients and investigators will be blinded to treatment. The Trial treatment will be a tablet formulation.

This Trial involves 11 clinic visits and 7 follow up telephone calls to reduce the burden of additional travel to the patients.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrolment:

1. The patient has a definitive diagnosis of Wolfram syndrome, as determined by the following:

   A) Documented diabetes mellitus diagnosed under 16 completed years according to WHO or ADA criteria plus documented optic atrophy diagnosed under 16 completed years

   AND B) Documented functionally relevant mutations on one or both alleles of the WFS1 gene based on historical test results (if available) or from a qualified laboratory at screening.
2. The patient is aged 6 years or older and weighing at least 20kg.
3. The patient's visual acuity assessed as either the right eye or left eye having a LogMAR score of 1.6 or better on an ETDRS chart, with or without corrected vision.
4. Written informed consent (and assent as required).
5. Females of child bearing potential will only be included after a negative highly sensitive urine pregnancy test. If sexually active, they must agree to use a highly effective contraception measure and to pregnancy testing at each clinic follow up visit- see 4.1.1 for further information.
6. Sexually active men with a female partner of childbearing potential must agree to the use of condoms and the use of a highly effective method of contraception by the female partner
7. Patient willing and able to meet all protocol defined visits for the duration of the Trial

Pregnancy

Adequate counselling must be given to all female patients of childbearing potential regarding the risks associated with Sodium Valproate use in pregnancy because of the potential teratogenic risk to the foetus. In the UK, Treat Wolfram protocol will be following the Valproate Pregnancy Prevention programme as per UK standard practice. Other countries will follow their local procedures as dictated by their local competent authority.

Female patients who have started their periods but are not sexually active will be given contraception advice. If under 16 years, the advice will be given to the patient and their parents or carers.

In line with Clinical Trial Facilitation Group Guidance, a woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Due to the potential teratogenic risk to the foetus, all women of childbearing potential (WOCBP) must use a highly effective method of contraception, without interruption during the entire duration of IMP treatment. A highly effective method of contraception according to the Clinical Trial facilitation Group guidance includes methods that can achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

* combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:

  * Oral
  * Intravaginal
  * Transdermal
* progestogen-only hormonal contraception associated with inhibition of ovulation:

  * Oral
  * Injectable
  * Implantable 1
* intrauterine device (IUD) 1
* intrauterine hormone-releasing system ( IUS) 1
* bilateral tubal occlusion 1
* vasectomised partner 1, 2
* sexual abstinence 3

  1. Contraception methods that in the context of this guidance are considered to have low user dependency.
  2. Vasectomised partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomised partner has received medical assessment of the surgical success.
  3. In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject.

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for this Trial:

1. The patient has clinically significant non-Wolfram related CNS involvement which is judged by the Investigator to be likely to interfere with the accurate administration and interpretation of protocol assessments.
2. The patient has a diagnosis of a mitochondrial myopathy
3. The patient has active liver disease, has a personal or family history of liver dysfunction related to known genetic disorders, or patient has porphyria.
4. The patient has received treatment with any investigational drug within the 30 days prior to Trial entry.
5. The patient is currently taking sodium valproate; or has a known hypersensitivity to sodium valproate or its excipients.
6. Any other acute or chronic medical, psychiatric, social situation or laboratory result that, based on investigator's judgment, would jeopardize patient safety during trial participation, cause inability to comply with the protocol, or affect the Trial outcome.
7. The patient is currently breastfeeding.
8. The patient has Known urea cycle disorders.
9. The patient has one of the following disorders: Lactose intolerance, the Lapp lactase deficiency, or glucose- galactose malabsorption.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Visual acuity (VA) | 36 months
  Visual acuity (VA) is measured on the logMAR scale by sight tests in clinic using Early treatment diabetic retinopathy study (ETDRS) charts. Values are taken for each eye separately, both uncorrected, and corrected with glasses or contact lenses, and can range from 0, which represents perfect vision i.e. 20/20 (values of -0.1 and -0.2 are also possible representing better than perfect vision), to +2 which represents near blindness i.e. 20/2000. Increases in logMAR represent deterioration.

SECONDARY OUTCOMES:
Safety - adverse events | 37 months
  measured by adverse events frequency, type and grade according to CTCAE v4
Tolerability - highest treatment dose | 36 months
  measured by dose achieved
Tolerability - duration of treatment | 36 months
  measured by days of treatment
Tolerability - dosing modifcation | 36 months
  measured by treatment-related dose reductions and discontinuations
Pons Volume | 37 months (+/- 6 months)
  a surrogate marker for neurodegeneration, measured and recorded in mm3 by standardised analysis of MRI images of the Pons, and brain substructure volumes.
Brainstem volume | 37 months (+/- 6 months)
  measured by MRI as with Pons Volume
Retinal nerve thickness | 37 months
  measured by Optical Coherence Tomography
Colour vision | 37 months
  measured by Hardy Rand and Rittler test
Visual fields | 37 months
  measured by the local centre standard process (the same technique must be used throughout the patient participation to the study)
Data on cataracts | 37 months
  measured by incidence and frequency of cataracts
Afferent pupillary defects | 37 months
  measured by incidence and frequency of afferent pupillary defects. Afferent pupillary defects are recorded as present or absent.
Strabismus | 37 months
  measured by incidence and frequency of strabismus. Presence or absence of strabismus will be recorded. Strabismus will also be graded for type and size.
Nystagmus | 37 months
  measured by incidence and frequency of nystagmus. Presence or absence of nystagmus will be recorded. Nystagmus will also be graded for size, amplitude and direction.
Visual evoked potentials | 37 months
  measured by changes in visual evoked potentials (if available)
Sleep - sleeping habits parent report for patients under 18 years | 37 months
  measured by the Sleep-related Breathing disorder scale extracted from the Pediatric Sleep Questionnaire (PSQ) Parent Questionnaire 2014. This report is a Parent Report for patients under 18. This questionnaire records usual sleep habits.
Sleep - sleeping habits, self-report | 37 months
  measured by the Pittsburg Sleep Quality Index (PSQI) Self-Report. This questionnaire is completed by the patient. This questionnaire records usual sleep habits during the past month.
Balance | 37 months
  measured by Mini-BESTest
Hearing | 37 months
  measured by pure tone audiometry
Wolfram Unified Rating Scale | 37 months
  Wolfram Unified Rating Scale (WURS). Assessments are performed in five areas (physical; seizure; behavioral; capability and clinical) by scoring listed items 0-2, 0-3, 0-4, 0-5 or 0-6 depending on the scale. Totals for each category are recorded and the WURS total, summing physical and behavioral categories, is also recorded. A low score would be considered a better outcome in all areas apart from capability where a high score would be considered a better outcome. A Wolfram Syndrome history is also recorded detailing incidence and onset of listed symptoms.
Mood | 36 months
  measured by Kidscreen for patients aged 8-18 or the Hospital Axiety and Depression Scale (HADS) for adult patients. Kidscreen records the patients mood and feeling in 5 areas (physical activities and health; general mood and feelings about self; family and free time; friends; school and learning). HADS records how the patient has been feeling over the past week by scoring feelings relating to anxiety or depression. A total score for Anxiety and a total score for depression is recorded. A score of 0-7 = normal; 8-10 = borderline abnormal (borderline case) and 11-21 = abnormal (case).
Quality of life - PedsQL | 37 months
  measured by PedsQL questionnaire (pediatric quality of life inventory) for paediatric patients. PedsQL 8-12 and PedsQL 13-18 and respective parent reports. PedsQL records how much of a problem each situation causes the patient; each situation is scored from 0 (never a problem) to 4 (always a problem). A score of 0 would be considered a better outcome.
Quality of life - ICIQ-FLUTS | 37 months
  measured by the ICIQ-FLUTS questionnaire: ICIQ-FLUTS (adult females), ICIQ-MLUTS (adult males), or ICIQ-CLUTS (children and caregiver forms). This questionnaire records urinary symptoms in three categories (filling, voiding and incontinence) from 0-4 and how much each symptom bothers the patient from 0 (not at all) to 10 (a great deal). Scores for each category are totalled. Low scores would be considered a better outcome.
Quality of life - VQoL_C/ YP | 37 months
  measured by the vision related quality of life questionnaire for children and for young people. This questionnaire records how patients feel about their eyesight in relation to the listed statements. Each statement is scored from 1 (not at all true) to 4 (completely true). The score denoting a better outcome is dependent on the question.
Quality of life - VFQ-25 | 37 months
  measured by the National Eye Institute Visual Function Questionnaire 25 (VFQ-25). This questionnaire records information in three categories. Questions in the general health and vision category are scored 1-5 or 6 and a low score would be considered a better outcome. Questions in the difficulty with activities category are scored 1 (no difficulty at all) to 6 (stopped doing this for other reasons or not interested in doing this); a low score would be considered a better outcome. Questions in the vision problems category are scored 1 (all of the time) to 5 (none of the time); a high score would be considered a better outcome.
Pancreatic beta cell reserve - glycated haemoglobin or equivalent | 37 months
  measured by percentage glycated haemoglobin or equivalent

OTHER OUTCOMES:
PBMC biomarker 1 | 37 months
  PBMC biomarker assay (p21cip1) (first measure) - assessing changes in patient during sodium valproate treatment and association with clinical outcome of treatment.
Genetic variations | 37 months
  Genetic variations associated with response to sodium valproate.
Gene expression changes | 37 months
  Gene expression changes associated with response to sodium valproate (including adverse effects)
Fractional anisotropy of the optic nerves | 37 months
  measured using Diffusion Tensor Imaging (DTI) on MRI
Global and regional brain volume measurements | 37 months
  to assess atrophy of brain structures by MRI
Change in Urodynamic function - 1st measure | 37 months
  measured by a primary micturition assessment for both day time and night time symptoms, as well as bowel assessment and the measurement of urinary flow rates upon void.
Change in Urodynamic function - 2nd measure | 37 months
  measured by the International Consultation on Incontinence Questionnaires (ICIQ) for Lower Urinary Tract Symptoms (LUTS), which evaluate lower urinary tract symptoms and impact on quality of life through patient reported outcome measures. Five versions of the ICIQ, each with 12 items, are used in the trial as follows: ICIQ-CLUTS - children up to the age of 18, 2 versions: one for children and one for parents/carers.
  ICIQ-FLUTS - adult females ICIQ-CLUTS - adult males
PMBC - Biomarker 2 | 37 months
  Lactate dehydrogenase (LDH) assay (second measure) - assessing changes in patient during sodium valproate treatment and association with clinical outcome of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Barrett, PhD, MB, BS, Principal Investigator — University of Birmingham
Locations (6):
- France (2):
  - CHU de Montpellier, Hopital Gui de Chauliac, Montpellier
  - Hôpital Européen Georges-Pompidou, Paris
- Medical University of Lodz, Lodz, Poland
- Unidad de Gestión Clínica Almería Periferia. Distrito Sanitario Almería, Almería, Spain
- United Kingdom (2):
  - University Hospitals Birmingham, Birmingham
  - Birmingham Women's and Children's Hospital, Birmingham

IPD SHARING:
Plan to Share IPD: No
No prior plans. CRCTU's data sharing policy - available here https://www.birmingham.ac.uk/research/crctu/data-sharing-policy.aspx - to be followed in the event of any plan to share.

REFERENCES:
- [Derived] Dias RP, Brock K, Hu K, Gupta R, Martin U, Peet A, Wilson M, Yu-Wai-Man P, Wright B, Mollan S, Kulkarni A, Meunier I, Billingham L, Nagy Z, Rose H, Koks S, Zatyka M, Astuti D, Lynch T, Morrison KE, Barton D, Cronier S, Malpass R, Evans R, Malhi A, Takhar P, Lamb A, Esteban-Bueno G, Mlynarski W, Orssaud C, Roubertie A, Homer V, Barrett T. Sodium valproate, a potential repurposed treatment for the neurodegeneration in Wolfram syndrome (TREATWOLFRAM): trial protocol for a pivotal multicentre, randomised double-blind controlled trial. BMJ Open. 2025 Feb 26;15(2):e091495. doi: 10.1136/bmjopen-2024-091495. PMID 40010822